CLINICAL TRIAL: NCT05715190
Title: Development and Feasibility of a Nurse-led Person-centered Education Program on Percentage Reduction of Psoriasis in Persons With Psoriasis: a Pilot Study
Brief Title: Development and Feasibility of a Nurse-led Person-centered Education Program
Acronym: PsoEd
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: School of Health Sciences Geneva (Other)
Collaborators: University of Lausanne Hospitals (Other); University of Lausanne (Other)
Responsible Party: Principal Investigator, Sebastian Probst, Full Professor of Tissue Viability and Wound Care, School of Health Sciences Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Psoriasis
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Self-Management; Behavior; Patient Empowerment
Keywords: patient education; self management; behavior change
MeSH Terms: conditions — Behavior; Patient Participation | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- nurse-led education (Other)
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Visiting the medical psoriasis outpatient clinic. Receiving a medical consultation, phototherapy and methotrexate treatment. Psoriasis plaque measurement, psoriasis care and questionnaires will be provided by the institute's nurses. After baseline data collection (T0) and random allocation to the intervention group, this usual care will be enhanced by a multidisciplinary nurse-led educational program

SUMMARY:
Background Psoriasis is a chronic inflammatory skin disease causing reduced quality of life. Psoriasis patients are often insufficiently informed about their disease with its treatment possibilities leading to non-adherence of treatment resulting in unsatisfactory patient outcomes. We therefore propose to develop an educational intervention for psoriasis patients; evaluate the feasibility of implementing it in a nurse-led psoriasis-outpatient clinic and compare the psoriasis percentage reduction, quality of life, health literacy and patient benefit, between patients receiving this educational intervention and those receiving standard care.

Method/Design We first will develop an evidence-based educational intervention in collaboration with an expert panel and second will conduct a quasi experimental feasibility study in a psoriasis outpatient clinic in Western Switzerland. Twenty four eligible patients with psoriasis will receive a multidisciplinary education, for 6 weeks. Data will be analyzed using R conducting linear models allowing us to assess the impact of the intervention on psoriasis reduction and other secondary outcomes of interest, once controlled for reliable socio-economic cofounding factors.

Discussion This trial will investigate the feasibility of the elaborated nurse-led education and the planed randomized controlled trial. In this study, we will elaborate and provide an informational brochure with information concerning psoriasis in addition to a nurse-led oral educational program in addition to medical standard care. We expect that this nurse-led person-centered intervention will contribute to enhanced education with a higher functioning, better self-efficacy and improved quality of life, better disease knowledge with a better adherence to the medication protocol. The results will further inform the final design of a subsequent large-scale randomized controlled trial, which will examine the effectiveness of this educational intervention. Additionally, through this study the role of the nursing profession and its research will be strengthened in assuring that the voice of individuals, families and communities are incorporated into design and operations of clinical health systems by eliminating gaps and disparities in health care.

DETAILED DESCRIPTION:
1. Introduction 1.1. Background and rationale Psoriasis is a systemic, immune-mediated disorder, characterized by inflammatory skin and joint manifestations that affects patient's quality of life, especially on a psychological, body aesthetic and social level, and therefore can impair not only their treatment adherence and sustainability of treatment but also patient-health care professional relationships. The psoriasis prevalence in adults in Europe ranges from 2% to 3%. If these findings are applied to the Swiss context it would mean that there are an estimated 180'000 persons suffering from psoriasis in Switzerland. The incidence increases with age making psoriasis a global health problem. Psoriasis can manifest in many different forms and is classified based on the severity of the disease into mild, moderate and severe. It is a chronic and recurrent disease being visible mostly on skin, which is characterized by alternating phases of outbreaks and remissions and whose evolution can vary greatly from one individual to another. Regardless of the severity, this chronic skin disease requires a long-term treatment strategy. Due to the visibility of lesions in patients and the inadequate understanding of this disease in public, individuals with psoriasis often suffer from stigma in their daily lives, which has adverse effects on their self-efficacy, mental health, quality of life, and therapeutic responses. A systematic review and meta-analysis by Xiao et al. show that for individuals suffering from psoriasis there are a variety of psychological intervention methods that are widely applied nowadays, among which cognitive behavioral therapy is the most recognized in the field. Cognitive behavioral therapy can reduce the stigma and confusion surrounding affective and anxiety responses to the disease, and it may improve psoriasis severity by inhibiting the inflammation associated with depression and anxiety. Consequences of stigmatization are low self-efficacy. Self-efficacy refers to an individual's self-perceived ability to act effectively in a variety of situations enhancing their activities of daily living. It is an important factor that influences the individual's ability to self-manage symptoms of their chronic diseases. Self-efficacy plays an important role in determining whether self-care actions are initiated, how much effort is exerted, and how long the effort is sustained in the face of obstacles and failures. Evidence demonstrates that if individuals with high self-efficacy in coping with their chronic diseases reflect a perceived ability to manage challenges related to their diseases and a sense of control over their lives. Self-efficacy in patients with psoriasis can be enhanced by education, acquiring coping skills through shared experiences or psychological support systems. Hence, psoriasis is a burden not only on the affected persons themselves, causing suffering and requiring lifelong management and treatments, but also on their close relatives and on society as a whole.

The care of patients with psoriasis has become, due to its complex chronic condition and course of disease, a specialty on its own. Traditionally, the therapeutic approach to the management of psoriasis is a multifaceted mostly medical approach determined by the type, the severity of the psoriasis, and the area of skin affected. Even though the etiology is not yet fully understood, traditionally, medical treatment options to decrease disease activity and improve symptoms are multifaceted including topical application of creams, phototherapy and/or systemic therapy. Topical treatment is mainly for mild or moderate psoriasis. This treatment includes ointments such as calcipotriol, calcineurin inhibitors, tretinoin, glucocorticoid, medicated bath with diastase or herbal extracts, and phototherapy. Phototherapy is an effective, safe, and accessible treatment without incurring any systemic side effects and can be combined with biologic agents for the treatment of more severe psoriasis. The systemic treatment involves conventional and newer oral or injectable systemic agents and biologics such as immune inhibitors, immune modulators or tumor necrosis factor α antagonists. Evidence reports an association between psoriasis severity and metabolic comorbidities, anxiety, depression, smoking, and alcohol abuse. An early diagnosis of these associated diseases, the implementation of treatment and adoption of healthy lifestyle are important in addition to the treatment of psoriasis symptoms to improve the prognosis.

In psoriasis patients, the level of knowledge about the pathogenesis and treatment of the disease has been shown to be insufficient. Evidence demonstrates that after six months a weekly two hours-educative session providing information on different aspects of psoriasis - including genetics, mechanisms, precipitating factors, course of the disease, preventive measures, co-morbidities, daily care of skin and treatment options, as well as psycho-educational guidance - can improve patient knowledge, and provide better coping strategies with the disease and better attitude towards therapy. A reduction of the psoriasis severity was reported by Bostoen and colleagues. They provided a physician driven education program about stress-reduction techniques with a 12-week education program (2h sessions twice a week), observing a reduction of disease severity and an improvement of quality of life, physical activity and depression status. These results are confirmed by Bubak's et al. prospective controlled study with 53 participants (24 IG, 29 CG), showing an increase in knowledge, self-expertise about the disease and amelioration of general health when participating in an educational program consisting in two 2h-workshops dealing with details on the etiology, pathogenesis, comorbidities, treatment options, nutrition, exercise, and addictions compared to usual care. However, there were no positive short-term effects seen on the quality of life and therapy adherence. A more recent study by Jendoubi and colleagues with 142 patients demonstrate that a standardized physician-led education program consisting of five sessions over 3 months improves patient knowledge and satisfaction but has no positive effect on quality of life of patients. Moreover, the results show that the program did not improve disease severity as well, which is in contradiction with the study of Bostoen and colleagues. Similarly, a randomized controlled trial including 64 psoriasis patients show no differences in psoriasis severity in participants attending a physician-led educational program consisting of 2-h sessions twice a week for 9 weeks versus the control group (IG: 5/46 [35.7%] vs.CG: 5/16 [31.3%]; p = 1.000). Hence, an educative program can allow to improve patient knowledge and satisfaction, but inconsistencies remain concerning its impact on the evolution of psoriasis severity and quality of life. Further studies are needed to optimize education programs improving disease severity and quality of life and how the benefits of such programs will evolve on the long-term needs also to be clarified.

Evidence reports that 26.6% of patients have low health literacy (HL) which is a higher percentage than the one observed for other chronic conditions. Health literacy is defined as knowledge of health, healthcare and health systems as well as processing and using information in various formats in relation to health and healthcare; and the ability to maintain health through self-management and working in partnerships with health providers. Low HL is associated with lower education, decreased communication with health care professionals, decreased ability to self-care, and higher psoriasis severity. High HL is a predictor of higher quality of life, self-efficacy, knowledge and reduced psoriasis severity. HL is therefore an important factor that may influence adherence to therapy and clinical outcomes in psoriasis patients. A cross-sectional study investigated the association between HL and psoriasis education from health care professionals in a cohort of 825 psoriasis patients using a 3 week-program (Climate Helio Therapy). Patients following the three-week program had a higher HL score (Cohen's effect size: 0.24 to 0.44), higher self-management and more psoriasis knowledge compared to participants who did not follow this program. However, this study didn't investigate the effectiveness of this program on psoriasis severity.

Nurses play an important and critical role in healthcare. The participation of nurses in comprehensive disease management is in countries such as the UK are well established. In Switzerland, this is slowly evolving, even though specialized nurses could take over more substantial aspects of patient care. Even though the nursing role is complementary to the one of a physician by advocating for health promotion, educate patients and the public on the prevention of illness, provide care and assist in cure, participate in rehabilitation, and provide support. This means that nurses have the opportunity to play a key role in transforming the health care system to create a more accessible, high-quality, and value-driven environment for patients. However, nowadays this role is inconsistently reported and is still poorly implemented in dermatology settings. In the field of wound care, this role is more established because nurses developed nurse-led wound clinics for complex wounds focusing mainly on education. Different modalities of patient education for example in the care of patients with venous leg ulcers have been reported including individual sessions, group sessions, telephone calls, web app based, audio-visual based, information leaflet or brochure. Evidence demonstrates that the use of various modalities may improve learning outcomes. Supporting information such as audiovisual or written content is important as people retain only a small amount of information from consultations. The majority of the education programs described above in psoriasis population are based on individual or group sessions. Only one pilot randomized controlled trial by Ersser and colleagues uses audio-visual, written materials and telephone calls in addition to group sessions, and another uses web app based education alone. However, research is needed to define the most appropriate model of nurse-led education program and to evaluate its effect on disease severity and quality of life. Therefore, we seek to develop a nurse-led educational intervention for psoriasis patients using selected educational modalities, evaluate its feasibility in clinical practice, and measure its impact on psoriasis severity in regards to quality of life, health literacy, and patient benefit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cutaneous psoriasis, regardless of the stage of the disease and treatment type (systemic and/or topic, and/or puva therapy)
* Age over 18 years
* Proficiency in the French language

Exclusion Criteria:

* Valid informed consent is not or cannot be given
* Patients unable to follow the 6-session therapeutic education program
* Patients currently engaged in any other therapeutic education program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-05-28 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
percentage reduction of psoriasi | 6 weeks
  percentage reduction of psoriasis using the PASI (Psoriasis Area and Severity Index) score. The intensity of redness, thickness, and scaling of the psoriasis is assessed as none (0), mild (1), moderate (2), severe (3), or very severe (4).

SECONDARY OUTCOMES:
Health Literacy | 6 weeks
  French version of the Health Literacy Survey European Questionnaire (HLS-EU-Q). scoring: 0 represented the lowest health literacy and 50 the highest health literacy
Patient benefit | 6 weeks
  patient benefit index short form (PBI-S) identifying patient needs by measuring the patient-relevant benefit of treatment, Patients with PBI-S ≥ 1 are considered having at least minimum patient-relevant treatment benefit
Life Quality Index | 6 weeks
  French version of the Dermatology Life Quality Index (DLQI) questionnaire
Psoriasis severity | 6 weeks
  French version of the self-administered psoriasis area and severity index (SAPASI)
Medication knowledge | 6 weeks
  standardized medication knowledge questionnaireincluding 11 questions with response categories being dichotomous (correct/not correct).
Knowledge of psoriasis | 6 weeks
  French version of the Psoriasis knowledge questionnaire (PKQ)
Self-management of the disease | 6 weeks
  French version of the Self-management efficacy questionnaire in psoriasis (SMEQ-PSO)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian E Probst, Prof, Principal Investigator — University of Applied Sciences and Arts Western Switzerland
Locations (1):
- Centre hospitalier universitaire vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
Open data source, Yareta